CLINICAL TRIAL: NCT01917214
Title: Patterns Of Care Among Australian Cohort Of Patients With Advanced Rrc Receiving Sutent
Brief Title: A Retrospective Real World Analysis Of Sutent In Patients With Metastatic Renal Cell Carcinoma In Community And Academic Centers To Assess The Impact Of Dose Variation On Duration Of Response And Overall Survival
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181210
Record Dates: First submitted 2013-07-25; First posted 2013-08-06 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Interventional Study
  Interventions: Other: Sutent: Observational Study

INTERVENTIONS:
Other: Sutent: Observational Study — Sutent oral therapy

SUMMARY:
This is a retrospective, non-interventional study which looks at the cohort of Renal Cell Carcinoma patients in a real life clinical setting and analyses into factors why these patients have been surviving for as long as 3-5 years unlike Clinical study where the survival is around 2 years.

The factors which will be analysed include patient characteristics, dosage and adverse event management and tries to correlate these factors with survival.

DETAILED DESCRIPTION:
A single cohort of 200 patients who are diagnosed with metastatic renal cell carcinoma prior to 1st Jan 2012, and are seen by the medical oncologist at the centers involved with BIOGRID and its affiliated registries. Patients will be identified from the first date of their consultation with the medical oncologist and captured in the electronic database. Consent to use datasets has already been obtained from participating research institutes and hospitals IRB/Ethics Committees

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Male or female
* Metastatic renal cell cancer
* First presentation with metastatic disease prior to 1st Jan 2012 since 2006, i.e. between 1st Jan 2006 to 31st Dec 2011

Exclusion Criteria:

* No referral to medical oncologist
* No record available in electronic database

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are diagnosed with metastatic renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181210&StudyName=A%20Retrospective%20Real%20World%20Analysis%20Of%20Sutent%20In%20Patients%20With%20Metastatic%20Renal%20Cell%20Carcinoma%20In%20Community%20And%20Academic%20Centers%20To%20As

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants diagnosed with mRCC who received either systemic therapy (Sutent [sunitinib malate] 25 milligram [mg], 37.5 mg or 50 mg or other systemic drugs [like bevacizumab, everolimus, pazopanib, sorafenib, temsirolimus]) OR best supportive care (BSC) as first line of treatment between 1 January 2006 and 31 December 2011 were observed retrospectively.
Period: Overall Study
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Started | 212
Completed | 212
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included participants diagnosed with metastatic renal cell carcinoma (mRCC) during the time period between 1 January 2006 and 31 December 2011.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 212
Age, Continuous [Median (Full Range); unit: years] — Age data was available for only 211 participants because 1 participant did not have date of diagnosis captured in the database and hence was excluded from the median age calculation.
  years | 60.73 [28.21 to 97.26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 [30.60 to 97.26]
  Male | 153 [28.21 to 89.08]

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) From Initiation of Sutent Therapy
Description: PFS was defined as the time from initiation of Sutent (sunitinib malate) to first documentation of tumor progression or to death due to any cause, whichever occurred first. Time to treatment failure was used as a surrogate for PFS as PFS could not be determined due to retrospective nature of this study.
Time Frame: From initiation of treatment up to 72 months
Population: Time to treatment failure (given in outcome measure 4) was used as a surrogate for PFS due to the lack of consistent regular restaging scans in clinical practice.
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Sutent Therapy: Participants diagnosed with mRCC who received systemic therapy with Sutent (sunitinib malate) 25 mg, 37.5 mg or 50 mg as first line of treatment between 1 January 2006 and 31 December 2011 were observed retrospectively.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort: Sutent Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate - Percentage of Participants With Objective Response From Initiation of Sutent Therapy
Description: Percentage of participants with objective response based on assessment of complete response (CR) or partial response (PR) as per clinical and radiological documentation in clinical notes. CR was defined as complete resolution of all visible disease, whereas PR was defined as partial reduction in size of visible disease.
Time Frame: From initiation of treatment up to 72 months
Population: Participants diagnosed with mRCC during the time period between 1 January 2006 and 31 December 2011 and received Sutent as a first-line therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort: Sutent Therapy
Number analyzed (Participants) | 125
percentage of participants | 30.4

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was the duration from diagnosis of disease to death. Overall survival was compared for those who had received best supportive care to those who received Sutent as first-line therapy.
Time Frame: From diagnosis until death (up to 72 months)
Population: Participants diagnosed with mRCC during time period between 1 January 2006 and 31 December 2011 and received Sutent or Best Supportive Care as a first-line therapy. Here, "N" (number of participants analyzed)=participants who were evaluable for this outcome measure. "n"=participants who were evaluable for this measure for each specified treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- mRCC Cohort: Sutent Therapy and BSC: Participants diagnosed with mRCC who received systemic therapy with Sutent (sunitinib malate) 25 mg, 37.5 mg or 50 mg OR best supportive care (BSC) as first line of treatment between 1 January 2006 and 31 December 2011 were observed retrospectively.
Arm/Group | mRCC Cohort: Sutent Therapy and BSC
Number analyzed (Participants) | 153
months
  Sutent (n=119) | 27.63 [18.88 to 34.97]
  Best Supportive Care (n=34) | 7.90 [2.86 to 31.48]
Statistical Analysis 1: Comparison: mRCC Cohort: Sutent Therapy and BSC; Test type: Superiority or Other; p = 0.0308, Log Rank

4. Secondary Outcome: Time to Treatment Failure From Initiation of Sutent Therapy
Description: Time to treatment failure was defined as the time from initiation of study treatment to the date of the first documentation of Progressive Disease (PD), symptomatic deterioration, death due to any cause, or discontinuation of treatment due to AE, refusal or other reason. PD was defined as an increase in visible disease.
Time Frame: From initiation of treatment up to 72 months
Population: Participants diagnosed with mRCC during the time period between 1 January 2006 and 31 December 2011 and received Sutent as a first-line therapy. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort: Sutent Therapy
Number analyzed (Participants) | 102
months | 8.95 [7.07 to 10.39]

5. Secondary Outcome: Correlation of Dosage and Number of Participants With CR (Complete Response), PR (Partial Response), SD (Stable Disease) and PD (Progressive Disease) From Initiation of Sutent Therapy
Description: Number of participants with CR, PR, SD and PD responses assessed as per clinical and radiological documentation in clinical notes for different Sutent doses were reported. CR was defined as complete resolution of all visible disease, PR was defined as partial reduction in size of visible disease, SD was defined as no change in size of visible disease, and PD was defined as an increase in visible disease. Here "other" refers to Sutent 12.5 mg.
Time Frame: From initiation of treatment up to 72 months
Population: Participants diagnosed with mRCC during the time period between 1 January 2006 and 31 December 2011 and received Sutent as a first-line therapy. Here, "n" signifies those participants who were evaluable for this measure for specified Sutent treatment.
Measure: Number; unit: participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort: Sutent Therapy
Number analyzed (Participants) | 125
participants
  Sutent 50 mg, CR (n=100) | 4 (0)
  Sutent 50 mg, PR (n=100) | 29
  Sutent 50 mg, SD (n=100) | 35
  Sutent 50 mg, PD (n=100) | 21
  Sutent 50 mg,Unknown (n=100) | 11
  Sutent 37.5 mg, CR (n=4) | 0
  Sutent 37.5 mg, PR (n=4) | 2
  Sutent 37.5 mg, SD (n=4) | 1
  Sutent 37.5 mg, PD (n=4) | 1
  Sutent 37.5 mg, Unknown (n=4) | 0
  Sutent 25 mg, CR (n=10) | 0
  Sutent 25 mg, PR (n=10) | 2
  Sutent 25 mg, SD (n=10) | 5
  Sutent 25 mg, PD (n=10) | 2
  Sutent 25 mg, Unknown (n=10) | 1
  Other, CR (n=1) | 0
  Other, PR (n=1) | 0
  Other, SD (n=1) | 0
  Other, PD (n=1) | 0
  Other, Unknown (n=1) | 1
  Unknown, CR (n=10) | 0
  Unknown, PR (n=10) | 1
  Unknown, SD (n=10) | 1
  Unknown, PD (n=10) | 3
  Unknown, Unknown (n=10) | 5

6. Secondary Outcome: Correlation of Duration and Number of Participants With CR (Complete Response), PR (Partial Response), SD (Stable Disease) and PD (Progressive Disease) From Initiation of Sutent Therapy
Description: Number of participants with CR, PR, SD and PD responses assessed as per clinical and radiological documentation in clinical notes for different durations of treatment with Sutent were reported. CR was defined as complete resolution of all visible disease, PR was defined as partial reduction in size of visible disease, SD was defined as no change in size of visible disease, and PD was defined as an increase in visible disease.
Time Frame: From initiation of treatment up to 72 months
Population: Participants diagnosed with mRCC during the time period between 1 January 2006 and 31 December 2011 and received Sutent as a first-line therapy. Here, "n" signifies those participants who were evaluable for this measure for specified treatment duration.
Measure: Number; unit: participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort: Sutent Therapy
Number analyzed (Participants) | 125
participants
  Less than (<) 3 months, CR (n=30) | 0 (0)
  <3 months, PR (n=30) | 2
  <3 months, SD (n=30) | 6
  <3 months, PD (n=30) | 16
  <3 months, Unknown (n=30) | 6
  3-6 months, CR (n=23) | 0
  3-6 months, PR (n=23) | 4
  3-6 months, SD (n=23) | 11
  3-6 months, PD (n=23) | 7
  3-6 months, Unknown (n=23) | 1
  6-12 months, CR (n=25) | 0
  6-12 months, PR (n=25) | 11
  6-12 months, SD (n=25) | 13
  6-12 months, PD (n=25) | 1
  6-12 months, Unknown (n=25) | 0
  12-24 months, CR (n=14) | 0
  12-24 months, PR (n=14) | 7
  12-24 months, SD (n=14) | 7
  12-24 months, PD (n=14) | 0
  12-24 months, Unknown (n=14) | 0
  Greater than (>) 24 months, CR (n=10) | 2
  >24 months, PR (n=10) | 5
  >24 months, SD (n=10) | 2
  >24 months, PD (n=10) | 0
  >24 months, Unknown (n=10) | 1
  Unknown, CR (n=23) | 2
  Unknown, PR (n=23) | 5
  Unknown, SD (n=23) | 3
  Unknown, PD (n=23) | 3
  Unknown, Unknown (n=23) | 10

ADVERSE EVENTS:
Description: Due to the retrospective nature of this study, adverse events (AEs) were not collected for this study.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Due to retrospective nature of this study, PFS could not be determined as restaging scans are not done on a consistent and regular basis in clinical practice. Time to treatment failure was used as a surrogate for PFS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days.

Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.